CLINICAL TRIAL: NCT05345080
Title: Phase 2 of the Houston "Breathe Easy" Healthy Homes-Based Model for Multifamily Rental Communities: Pragmatic Clinical Trial
Brief Title: Houston "Breathe Easy" Healthy Homes-Based Model for Multifamily Rental Communities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Baylor College of Medicine (Other)
Collaborators: Harris County Hospital District (Other Government); The University of Texas Health Science Center, Houston (Other); Oregon State University (Other)
Responsible Party: Principal Investigator, Winifred J. Hamilton, PhD, Associate Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-46145; TXHHU0043-18 (Other Grant/Funding Number: U.S. Department of Housing & Urban Development)
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Asthma; Respiratory Tract Disease; Lung Diseases; Sinusitis, Chronic
Keywords: asthma; environmental triggers; phone-based intervention; public housing; apartments
MeSH Terms: conditions — Asthma; Respiratory Tract Diseases; Lung Diseases; Sinusitis; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure-Reduction Intervention Group (Experimental): The exposure-reduction (intervention) group receives a phone-based telehealth visit, collection of self-report information from detailed health and exposure questionnaires, asthma education, assessment for allergies (optional), a customized asthma self-management plan and support developed using motivational interviewing methods, and a customized selection of supplies to help reduce key exposures likely exacerbating asthma symptoms.
  Interventions: Behavioral: Exposure-Reduction Intervention
- Phone-Call-Only Control Group (No Intervention): The phone-call-only (control) group provides self-reported information about health and environmental exposures. They receive follow-up phone calls every 6 weeks to maintain contact only. After exit, the phone-call-only (control) group receives assessment for allergies (optional) and the exposure-reduction intervention.

INTERVENTIONS:
Behavioral: Exposure-Reduction Intervention — The customized exposure-reduction intervention includes a phone-based telehealth visit, collection of self-report information from detailed health and exposure questionnaires, asthma education, assessment for allergies (optional), and a customized asthma self-management and exposure-reduction plan developed using motivational interviewing techniques, support, and exposure-reduction supplies.
  Arms: Exposure-Reduction Intervention Group

SUMMARY:
The primary purpose of this pragmatic randomized clinical trial is to examine whether the addition of a phone-based multicomponent environmental intervention customized for Houston public housing residents with asthma will result in statistically significant improvements in key measures of health, quality of life, and resilience.

DETAILED DESCRIPTION:
This is a pragmatic randomized clinical trial that examines the effectiveness of a clinically informed phone-based environmental intervention for improving asthma control in individuals living in selected Houston Housing Authority public housing communities. This study was initially designed as an in-home intervention but changed to a phone-based intervention, with drop-offs of supplies and other materials, because of the coronavirus pandemic. Both the control and intervention groups complete a comprehensive set of questionnaires by phone (or online or on paper), and wear a passive wristband collection device for seven days that measures exposure to 1,530 chemicals. Each enrollee is randomly assigned into one of the two groups after the baseline questionnaires are completed. The intervention ("exposure-reduction") group receives a telehealth visit, a customized Multicomponent Asthma Action Plan, multiple phone-based intervention visits and customized exposure-reduction supplies and materials, delivered to their porch, to implement the plan and support behavior change. The exposure-reduction group is encouraged to provide a blood sample to a local Harris Health laboratory for analysis of allergic and eosinophilic status. The control ("phone-call-only") group receives phone follow-up calls. Six months after the baseline assessment, both groups are reassessed at the exit visit. The phone-call-only group receives the exposure-reduction intervention after the exit visit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of poorly controlled asthma*
* Live in one of the selected public housing communities operated by the Houston Housing Authority
* No clear plan to move within the next 6 months
* Working telephone number
* Able to read and speak in English

  * Poorly controlled asthma defined as (1) has been diagnosed by a physician as having asthma in the past and currently has asthma; and (2) fulfills one or more of the following criteria of poorly controlled asthma: has had one or more emergency department visits or hospitalizations for asthma in the preceding year; has had asthma symptoms during the daytime at least two days in the past week; has been awoken at night by asthma symptoms one or more nights in the past week; or has used asthma rescue medication at least twice in the past week. These eligibility criteria effectively include two categories of asthma control as defined by the National Asthma Education and Prevention Program, (NAEPP) Third Expert Panel (EPR3) on the Diagnosis and Management of Asthma: "not well controlled" and "very poorly controlled" asthma.

Exclusion Criteria:

* Severe co-morbid conditions--such as a poorly controlled psychiatric illness or a condition requiring intense medical treatment--that could reasonably be expected to (1) confound the effects of this study's intervention or (2) make it unlikely that a participant could follow the treatment plan.
* A concurrent pulmonary study that could reasonably be expected to confound the effects of the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Asthma Control Test (ACT) Score | Measured at baseline and 6 months later
  The ACT is a validated 5-question scale assessing asthma control over the previous four weeks. Each question has five possible responses, from 1 (worst) to 5 (best). The total score ranges from 5 (worst control) to 25 (best control). In general, a total score of 19 or less suggests poor asthma control.
Change in Juniper Mini Asthma Quality of Life Questionnaire (MiniAQLQ) Score | Measured at baseline and 6 months later
  A validated 15-item questionnaire, with each question having seven possible answers score from 1 (worst) to 7 (best). Minimum total score is 15 (worst asthma quality of life). Maximum total score is 105 (best asthma quality of life). By design, an individual's score is reported as the mean (total score/15). Thus the possible mean reported score ranges from 1 (worst asthma quality of life) to 7 (best asthma quality of life).

SECONDARY OUTCOMES:
Change in Emergency Department (ED) Visits | Collected at baseline and 6 months later (for the preceding 6 months)
  The healthcare utilization questions were from the validated CDC-BRFSS Asthma Survey. For this outcome measure, patient responses to a question that asked "During the past 6 months, how many times to you visit an emergency room of urgent care center because of your asthma?" were used.

CONTACTS AND LOCATIONS:
Overall Officials: Winifred J Hamilton, PhD, SM, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant lab results and a progress note are posted in the participant's Harris Health electronic medical record (EMR). Low enrollment limits the usefulness of data sharing with other researchers at the individual level.